CLINICAL TRIAL: NCT03180320
Title: Effect of an Exercise-based Cardiac Rehabilitation Program 'Baduanjin-eight-silken-movement With Self-efficacy Building' for Patients With Chronic Heart Failure in Guangzhou, China (BESMILE-HF Study)
Brief Title: Baduanjin-eight-silken-movement With Self-efficacy Building for Patients With Chronic Heart Failure (BESMILE-HF Study)
Acronym: BESMILE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Weihui Lu, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2016-202-01
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure
Keywords: chronic heart failure; exercise-based cardiac rehabilitation; Baduanjin
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: Given the nature of the intervention, it is not possible to blind the patients and personnel involved in conducting the programs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BESMILE-HF group (Experimental): Throughout the study period, all participants will receive typical Western medications for chronic heart failure, according to national guidelines. In addition, patients will receive the BESMILE-HF program.
  Interventions: Behavioral: BESMILE-HF program; Drug: Usual medications
- Control (Other): Patients in the control group will receive only the usual medications, since patients typically do not receive exercise-based cardiac rehabilitation in this kind of setting.
  Interventions: Drug: Usual medications

INTERVENTIONS:
Behavioral: BESMILE-HF program — The following activities will be conducted as part of the BESMILE-HF program:
  1. Baduanjin exercise;
  2. evaluations of exercise capacity and clinical conditions;
  3. consultations on exercise prescription and management of symptoms/signs during exercise;
  4. education covering topics related to the CHF and exercise; and
  5. a series of adherence strategies.
  Arms: BESMILE-HF group
Drug: Usual medications — Throughout the study period, all participants will receive typical Western medications for chronic heart failure, according to national guidelines.

SUMMARY:
Chronic heart failure (CHF) is a major and growing public health problem and poses economic burden on the society. There is a need for a safe, equipment-free, low-cost, and easily implemented exercise-based cardiac rehabilitation program for CHF patients in China. Baduanjin exercise, translated as 'eight silken movements', is one of the most common forms of traditional Chinese exercise and it could have value to be integrated into a exercise-based cardiac rehabilitation program for CHF patients, together with education, evaluation and consultancy. Accordingly, the BESMILE-HF program applying the Baduanjin exercise as the central component, has been developed in Guangdong Provincial Hospital of Chinese Medicine which is one of the largest hospitals of Chinese medicine in China. This project is to evaluate the efficacy and acceptability of BESMILE-HF program in patients with CHF in China, and it will be based on a randomized controlled trial and a qualitative study.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or above
2. diagnosed with chronic heart failure
3. clinically stable as defined as symptoms and signs that have remained generally unchanged for at least 1 month
4. NYHA functional class II or III

Exclusion Criteria:

1. patients who have contraindications to cardiopulmonary test
2. patients who have contraindications to exercise training
3. Patients who have serious acute or chronic organic disease or mental disorders
4. history of cardiac surgery, cardiac resynchronization therapy, or intracardiac defibrillation within the previous 3 months;
5. history of cardiac arrest within 1 year;
6. history of peripartum cardiomyopathy, hyperthyroid heart disease, primary pulmonary hypertension;
7. inability to perform a bicycle stress test;
8. severe cognitive dysfunction precluding informed consent or understanding of exercise concepts;
9. current regular Baduanjin or current participation in a conventional cardiac rehabilitation program
10. current participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline peak VO2 (ml/kg/min) at 12 week | Baseline, 12 week
  Peak oxygen uptake
Change from baseline MLHFQ at 12 week | Baseline,12 week
  Minnesota Living with Heart Failure Questionnaire

SECONDARY OUTCOMES:
6MWT | Baseline, 4 week, 8 week, 12 week
  6-minute walking test
TGUG | Baseline, 4 week, 8 week, 12 week
  Timed get-up and-go
SEE-C | Baseline, 4 week, 8 week, 12 week
  Exercise Self-efficacy
MLHFQ | Baseline, 4 week, 8 week, 12 week
  Minnesota Living with Heart Failure Questionnaire
EQ-5D | Baseline, 4 week, 8 week, 12 week
  General quality of life
GRC | Baseline, 4 week, 8 week, 12 week
  Global Rating of Change
LVEDD (mm) | Baseline, 12 week
  Parameters from echocardiography: Dimensions and volumes
LA (mm) | Baseline, 12 week
  Parameters from echocardiography: Dimensions and volumes
LVEF (%) | Baseline, 12 week
  Parameters from echocardiography: Left ventricular systolic function
Global longitudinal strain 2D (%) | Baseline, 12 week
  Parameters from echocardiography: Left ventricular systolic function
E/A ratio | Baseline, 12 week
  Parameters from echocardiography: Left ventricular diastolic function
NT pro-BNP | Baseline, 12 week
  Prognostic biomarker from blood sample
hsCRP | Baseline, 12 week
  Inflammatory indicator from blood sample
Total score of Patient Health Questionnaire-9 (PHQ-9) | Baseline, 4 week, 8 week, 12 week
  The total score ranges from 0-27, the higher scores indicates worse outcomes
Total score of General Anxiety Disorder-7 (GAD-7) | Baseline, 4 week, 8 week, 12 week
  The total score ranges from 0-21, the higher scores indicates worse outcomes
Number of patients who has a increand 6% PeakVO2 | Baseline, 12 week
  Number of patients who has a increand 6% PeakVO2

OTHER OUTCOMES:
IPAQ | Baseline, 4 week, 8 week, 12 week
  International Physical Activity Questionnaire
Adverse events | Through study completion, an average of 12 weeks
  Safety assessment
MACEs | Through study completion, an average of 12 weeks
  Major acute cardiac events
SDANN Index | Baseline, 12 week
  Parameters from Holter 24-hour ECG
SDNN Index | Baseline, 12 week
  Parameters from Holter 24-hour ECG
All-caused mortality All-caused mortality | Through study completion, an average of 12 weeks
  All-caused mortality
All-caused hospitalization | Through study completion, an average of 12 weeks
  All-caused hospitalization
Heart failure hospitalizaiton | Through study completion, an average of 12 weeks
  Heart failure hospitalizaiton

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Lu, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine; Gaetano Marrone, Principal Investigator — Karolinska Institutet; Wei Jiang, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine; Zehuai Wen, Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun P, Cen H, Chen S, Chen X, Jiang W, Zhu H, Liu Y, Liu H, Lu W. Left atrial dysfunction can independently predict exercise capacity in patients with chronic heart failure who use beta-blockers. BMC Cardiovasc Disord. 2023 Mar 9;23(1):128. doi: 10.1186/s12872-023-03127-9. PMID 36894879
- [Derived] Chen X, Jiang W, Olson TP, Lundborg CS, Wen Z, Lu W, Marrone G. Feasibility and Preliminary Effects of the BESMILE-HF Program on Chronic Heart Failure Patients: A Pilot Randomized Controlled Trial. Front Cardiovasc Med. 2021 Jul 27;8:715207. doi: 10.3389/fcvm.2021.715207. eCollection 2021. PMID 34386535
- [Derived] Chen X, Jiang W, Lin X, Lundborg CS, Wen Z, Lu W, Marrone G. Effect of an exercise-based cardiac rehabilitation program "Baduanjin Eight-Silken-Movements with self-efficacy building" for heart failure (BESMILE-HF study): study protocol for a randomized controlled trial. Trials. 2018 Mar 1;19(1):150. doi: 10.1186/s13063-018-2531-9. PMID 29490680